CLINICAL TRIAL: NCT06694909
Title: Glutamate Modulation of tDCS Over Premotor Cortex Combined With Peripheral Nerve Stimulation Promoted Observation-execution-related Cortical Excitability and Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GMOTOPCCWPNSPOERCEAML
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Brain Stimulation; Peripheral Nerve Stimulation; Motor Observation; Cortical Excitability
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- tDCS + PNS with action observation (Experimental)
  Interventions: Device: tDCS + PNS without action observation
- sham tDCS + sham PNS with action observation (Experimental)
  Interventions: Device: sham tDCS + sham PNS with action observation
- tDCS + PNS without action observation (Experimental)
  Interventions: Device: sham tDCS + PNS with action observation
- sham tDCS + PNS with action observation (Active Comparator)
  Interventions: Device: tDCS + PNS with action observation
- tDCS + sham PNS with action observation (Active Comparator)
  Interventions: Device: tDCS + sham PNS with action observation

INTERVENTIONS:
Device: tDCS + PNS with action observation — tDCS: transcranial direct current stimulation; PNS: peripheral nerve stimulation
  Arms: sham tDCS + PNS with action observation
Device: sham tDCS + sham PNS with action observation — tDCS: transcranial direct current stimulation; PNS: peripheral nerve stimulation
  Arms: sham tDCS + sham PNS with action observation
Device: tDCS + PNS without action observation — tDCS: transcranial direct current stimulation; PNS: peripheral nerve stimulation
  Arms: tDCS + PNS with action observation
Device: sham tDCS + PNS with action observation — tDCS: transcranial direct current stimulation; PNS: peripheral nerve stimulation
  Arms: tDCS + PNS without action observation
Device: tDCS + sham PNS with action observation — tDCS: transcranial direct current stimulation; PNS: peripheral nerve stimulation
  Arms: tDCS + sham PNS with action observation

SUMMARY:
This study aimed to investigate whether concurrent tDCS over the PMC and PNS during action observation enhance observation-execution-related motor cortex excitability and improve motor performance, and to explore the underlying mechanism

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected-to-normal vision
* right-handed

Exclusion Criteria:

* pregnancy
* a history of epilepsy
* implanted medical devices
* history or presence of neurological, psychiatric or musculoskeletal disorders, other medical conditions, and left-handedness

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Motor-evoked potentials | Before interventions, and immediately after interventions
intracortical facilitation assessed by transcranial magnetic stimulation | Before interventions, and immediately after interventions
short-interval intracortical inhibition assessed by transcranial magnetic stimulation | Before interventions, and immediately after interventions
Reaction times of action execution blocks | immediately after interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, Haidian, China